CLINICAL TRIAL: NCT05586217
Title: Effects of Incentive Spirometry on Dyspnea and Chest Clearance in Asthmatic Patients During Seasonal Smog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/0332 Muhadsa Chaudhary
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Shortness of Breath
Keywords: Spirometry,Asthma,Dyspnea and Chest clearance
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive Spirometry (Experimental): 12 weeks, 1 session per week; each session took about 1 hour.
  Interventions: Other: INCENTIVE SPIROMETRY; Other: Active cycle of breathing
- Active Cycle of Breathing (Active Comparator): Breathing Control Deep Breathing Exercises or Thoracic Expansion Exercises Huffing or Forced Expiratory Technique (FET)
  Interventions: Other: Active cycle of breathing

INTERVENTIONS:
Other: INCENTIVE SPIROMETRY — * Sit up and hold the device.
  * Then Place the mouthpiece spirometer in mouth and make a good seal over the mouthpiece with lips.
  * Breathe out (exhale) normally.
  * Breathe in (inhale) slowly. A piece in the incentive spirometer will rise as you breathe in. And try to get this piece to rise as high as you can.
  * Usually, there is a marker placed by your doctor that tells you how big of a breath you should take.
  A smaller piece in the spirometer looks like a ball or disk.
  * Your goal should be to make sure this ball stays in the middle of the chamber while you breathe in.
  * If you breathe in too fast, the ball will shoot to the top.
  * If you breathe in too slowly, the ball will stay at the bottom. Hold your breath for 3 to 5 seconds. Then slowly exhale.
  Arms: Incentive Spirometry
Other: Active cycle of breathing — Breathe in and out gently through your nose if you can. If you cannot, breathe through your mouth instead. If you breathe out through your mouth, it's best to use breathing control with 'pursed lips breathing'. keep your shoulders relaxed.
  Try closing your eyes to help you to focus on your breathing and to relax. Breathing control should continue until the person feels ready to progress to the other stages in the cycle. Try to keep your chest and shoulders relaxed.
  At the end of the breath in, hold the air in your lungs for 2-3 seconds before breathing out. Breathe out gently and relaxed. Repeat 3 - 5 times. Sit up straight with chin tilted slightly up and mouth open.
  Take a slow deep breath to fill lungs about three quarters full. Hold breath for two or three seconds. Exhale forcefully, but slowly, in a continuous exhalation to move mucus from the smaller to the larger airways

SUMMARY:
EFFECTS OF INCENTIVE SPIROMETRY ON DYSPNEA AND CHEST CLEARANCE IN ASTHMATIC PATIENTS DURING SEASONAL SMOG

DETAILED DESCRIPTION:
Asthma is a serious and life threatening chronic respiratory disease that affects the quality of life of more than 23 million Americans- with exposure to air pollution. Air pollution can make asthma symptoms worse and trigger asthma attacks. Particle pollution can cause breathing problems. It's created when tiny bits of dust, dirt, smoke, soot, and other stuff hang in the air. The smaller the particles, the deeper they can get into the lungs and cause breath problems. Seasonal smog aggravates asthma, irritates the lungs, and makes it difficult to breathe. Long-term inflammation from breathing in too much ground-level ozone can permanently scar lung tissue. Smog with high levels of ozone is also particularly damaging for people with asthma. During seasonal smog asthma patients are more affected than normal people. Various consecutive treatments are used to treat the asthma patients for the improvement of quality of life. But at this check the effects of incentive spirometry on dyspnea and chest clearance in asthmatic patients.

This study will be randomized controlled trial. This study will be conducted in Ittefaq Hospital Lahore. Subjects meeting the predetermined inclusion and exclusion criteria. Sample size will be 44 including both male and female. QUESTIONNAIRE used as subjective measurements and ASHMA CONTROL TEST as objective measurement. Dyspnea-12 will be used to check the dyspnea severity in asthma patients and asthma control test will be used to check asthma severity during seasonal smog. Cough and sputum assessment questionnaire will be used to check effectiveness of chest clearance. Subjects of one group will be treated with active cycle of breathing and incentive spirometry and the other group will be treated with only spirometry. Each group will receive 12 treatment sessions with one treatment session per week and it will take less than 1 hour. Pre- treatment reading of dynpnea-12, cough and sputum assessment questionnaire and asthma control test will be recorded. And post-treatment readings will also be recorded.

Outcome variables will be dyspnea-12, incentive spirometry, cough and sputum assessment questionnaire and asthma control test. Most commonly used incentive spirometry to clear the dyspnea and chest clearance in asthma patients. Data will be analyzed on SPSS-25.

ELIGIBILITY:
Inclusion Criteria:

* Age group:30-45
* Patients of bronchial Asthma
* Patients who have difficulty in breathing

Exclusion Criteria:

* Age:<30 yrs->45 yrs
* Patients of COPD,Bronchiectasis,Pneumonia,Pulmonary TB or any other chronic lung disease.
* Patients of HTN, IHD, patients of fever or any other chronic disease

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-09-10 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Asthma Control test | 12 weeks
  In asthma control test we use spirometer to check out the respiratory functions.
Incentive Spirometry | 12 weeks
  An incentive spirometer is a handheld medical device that measures the volume of our breath.
  It helps our lungs recover after surgery or lung illness, keeping them active and free of fluid.

OTHER OUTCOMES:
Dyspnea-12 | 12 weeks
  in Dyspnea-12 we use spirometer to check out the dyspnea.
Cough and Sputum assessment questionnaire | 12 weeks
  in cough and sputum assessment questionnaire we use spirometer to check out the chest clearance.

CONTACTS AND LOCATIONS:
Overall Officials: sumera abdulhameed, MS, Principal Investigator — Riphah International University
Locations (1):
- Iettefaq hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No